CLINICAL TRIAL: NCT04826172
Title: A Randomized, Double-Blind, Placebo-Controlled, Exploratory Study on the Safety, Tolerability, and Pharmacodynamics of IMB-1018972 in Subjects With Angina Due to Obstructive Coronary Artery Disease
Brief Title: Exploratory Study on the Safety, Tolerability, and Pharmacodynamics of IMB-1018972 in Subjects With Angina Due to Obstructive Coronary Artery Disease (IMPROVE-Ischemia)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imbria Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMB101-006
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Ischemia; Coronary Artery Disease
MeSH Terms: conditions — Ischemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IMB-1018972 200mg (Experimental)
  Interventions: Drug: IMB-1018972
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMB-1018972 — Modified release (MR) oral tablet
  Arms: IMB-1018972 200mg
Drug: Placebo — Matching oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of IMB-1018972 in subjects with obstructive CAD and inducible ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of stable angina (CCS grading I-III) or anginal equivalent for ≥1 month prior to screening
* Ability to safely abstain from beta blockers for 48 hours prior to echo examinations in the opinion of the Investigator
* Preserved LV systolic function, defined as LVEF≥50% by any imaging modality
* Obstructive CAD and recent evidence of stress-induced myocardial ischemia

Exclusion Criteria:

* Women of childbearing potential or who are currently pregnant or breast-feeding
* Clinically indicated for coronary revascularization (PCI/CABG) at time of screening or clinically significant LMS or proximal LAD stenosis likely to warrant revascularization during the study period in the opinion of the investigator.
* Type 1 insulin dependent diabetes mellitus (IDDM)
* Presence of pacemaker, cardiac resynchronization therapy and/or implantable cardioverter defibrillator
* Severe or clinically significant valvular heart disease
* Clinically significant concurrent condition which could prevent the patient from performing any of the protocol-specified assessments, represent a safety concern if the patient participates in the trial or could confound trial assessments of safety or tolerability

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IMB-1018972 as measured by incidence and severity of treatment emergent AEs (including AEs leading to study drug discontinuation and AEs leading to death), as well as incidence of treatment emergent SAEs | Randomization through Week 10 Safety Follow-up

SECONDARY OUTCOMES:
Change in number of ischemic segments during hyperemia (ischemia defined as absolute MBF ≤2.0 ml/kg/min) as measured by adenosine stress 15O-H2O PET | Baseline through Week 8
  Ischemia score defined on the basis of absolute hyperemic MBF as: (1) MBF 2.0-2.3 ml/g/min; (2) 1.7- 2.0 ml/g/min; (3) MBF <1.7 ml/g/min
Change in total ischemia burden measured as ischemia score summed across all segments as measured by adenosine stress 15O-H2O PET | Baseline through Week 8
Change in inducible perfusion defect expressed as % of myocardium as measured by adenosine stress 15O-H2O PET | Baseline through Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Chair — Imbria Pharmaceuticals, Inc.
Locations (3):
- Imbria Investigational Site, Aarhus, Denmark
- Imbria Investigational Site, Turku, Finland
- Imbria Investigational Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided